CLINICAL TRIAL: NCT00268255
Title: Phase I/II Study of Induction Gefitinib and Concurrent Radiotherapy in Patients With Previously Untreated, Medically Inoperable Stage I or II Non-Small Cell Lung Cancer
Brief Title: Gefitinib and Radiation Therapy in Treating Patients With Inoperable Stage I or Stage II Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study never moved forward with accrual.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000447160; WSU-D-2820; WSU-HIC-100304M1F; ZENECA-1839US/0258
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma of Lung | interventions — Gefitinib; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gefitinib
Procedure: adjuvant therapy
Procedure: enzyme inhibitor therapy
Procedure: neoadjuvant therapy
Procedure: protein tyrosine kinase inhibitor therapy
Procedure: radiation therapy
Procedure: radiosensitization

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Gefitinib may make tumor cells more sensitive to radiation therapy. Giving gefitinib together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of radiation therapy when given together with gefitinib and to see how well they work in treating patients with inoperable stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity profile and maximum tolerated dose of radiotherapy when given in combination with gefitinib in patients with previously untreated, medically inoperable stage I or II non-small cell lung cancer. (Phase I)
* Determine the efficacy of gefitinib when given for 6 weeks prior to and concurrent with radiotherapy, in terms of objective response rate (partial and complete response), in these patients.

Secondary

* Determine the 3-month tumor response (complete and partial response) in patients treated with this regimen.
* Determine the 6-week response rate in patients treated with this regimen.
* Determine the local disease control rate (complete and partial response, stable disease) in patients treated with this regimen.
* Determine the local progression-free survival and disease-specific survival (cancer vs co-morbid disease) of patients treated with this regimen.
* Determine the pattern of failure (e.g., local, regional, or distant metastasis) in patients treated with this regimen.
* Determine the acute and late radiation toxic effects to organs at risk in patients treated with this regimen.
* Determine the safety profile of gefitinib in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of radiotherapy.

* Patients receive oral gefitinib once daily for 13 weeks. Patients also undergo radiotherapy 5 days a week for 7 weeks beginning at week 7. Patients continue to receive gefitinib alone after completion of radiotherapy in the absence of disease progression or unacceptable toxicity.

Cohorts of 6-10 patients receive escalating doses of radiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience acute dose-limiting toxicity.

* Phase II: Patients receive oral gefitinib as in phase I and radiotherapy at the MTD determined in phase I. After the completion of radiotherapy, patients continue to receive gefitinib in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A maximum of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)
* Any non-small cell histology allowed
* T1-3, N0* disease
* No metastatic disease
* Refused or ineligible for surgery
* Measurable disease, defined as lesion diameter ≤ 5 cm NOTE: *No evidence of N1 or N2 disease by positron emission tomography (PET) scan or any histological means (mediastinoscopy, thoracotomy, transbronchial, tracheal aspirations, or transesophageal aspiration by endoscopic ultrasound guidance

PATIENT CHARACTERISTICS:

Performance status

* Any performance status

Life expectancy

* At least 1 year

Hematopoietic

* No restrictions

Hepatic

* No restrictions

Renal

* Creatinine ≤ CTC grade 2

Pulmonary

* No clinically active interstitial lung disease
* Chronic, stable, asymptomatic radiographic changes allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No known severe hypersensitivity to gefitinib or any of the excipients of this product
* No other malignancy within the past 5 years except basal cell cancer or carcinoma in situ of the cervix
* No active or uncontrolled infection
* No uncontrolled systemic disease
* No psychiatric illness or other severe medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Radiotherapy

* No prior radiotherapy to the chest or mediastinum
* No concurrent elective nodal irradiation

Surgery

* Recovered from prior surgery
* No concurrent ophthalmic surgery

Other

* Recovered from all other prior anticancer therapy (alopecia allowed)
* More than 30 days since prior nonapproved or investigational agents
* No concurrent CYP3A4 inducers, including any of the following:
* Phenytoin
* Carbamazepine
* Barbiturates
* Rifampin
* Phenobarbital
* Hypericum perforatum (St. John's wort)
* No concurrent systemic retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T. Turrisi, MD, Study Chair — Barbara Ann Karmanos Cancer Institute